CLINICAL TRIAL: NCT06043895
Title: The Overall Surgical Time Comparison Between EpiFaith® CV and Conventional Syringe in Central Venous Catheterization
Brief Title: EpiFaith CV for Central Venous Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 202304082DIND
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Catheterization, Central Venous; Equipment Design; Patient Safety; Anesthesiology Devices Associated With Misadventures, Diagnostic and Monitoring Devices; Perioperative Care
Keywords: Central Venous Catheterization; Patient Safety; Visual Feedback; Anesthesiology; Clinical Skill
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The care providers (conducting physicians) and the research assistants who observe and record the results will know the assignments, while the participants and data analysts will not know the assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EpiFaith CV (Experimental): The conducting physicians in this group will use EpiFaith CV to localize the central vein and assess if there is arterial puncture
  Interventions: Device: EpiFaith CV
- Conventional (Active Comparator): The conducting physicians in this group will use Raulerson syringe to localize the central vein and assess if there is arterial puncture
  Interventions: Device: Conventional

INTERVENTIONS:
Device: EpiFaith CV — The conducting physician will localize the central vein using EpiFaith CV and assess if there is arterial puncture.
  Arms: EpiFaith CV
Device: Conventional — The conducting physician will localize the central vein using Raulerson syringe and assess if there is arterial puncture.
  Arms: Conventional

SUMMARY:
EpiFaith CV provides automatic aspiration and detection of arterial pressure as an alternative to manometry in central venous catheterization. The aim of the study is to evaluate if it may reduce operation time compared with conventional syringe.

DETAILED DESCRIPTION:
Central venous catheterization (CVC) is crucial in modern perioperative and intensive care. Keeping constant and stable negative pressure while advancing the needle had been issue for beginners. Recently, EpiFaith CV provides a new solution for CVC, which facilitates syringe control and precision during assessing vessels. It provides steady aspiration and detection of arterial pressure as an alternative to manometry without the need to disconnect nor more connections. The aim of the study is to evaluate if it may reduce operation time compared with conventional syringe.

ELIGIBILITY:
Inclusion Criteria (for participants):

* 18 years old and above
* Surgical patients who need to have a central venous catheter placed
* Informed and agree to participate in the study

Inclusion Criteria (for conducting physicians):

* Physicians with >100 central venous catheter placement experience, including attending physicians and senior residents

Exclusion Criteria (for participants):

* Patient refusal
* Puncture site skin lesions
* Uncorrected coagulation disorder
* Hemodynamic instability
* Not informed and consented to participate in research

Exclusion Criteria (for conducting physicians):

* Not informed and consented to participate in research

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The overall surgical time | 1 hour
  The time from needle insertion, aspiration of blood, assessment of vein or artery, insertion of guidewire, until removal of the needle

SECONDARY OUTCOMES:
Amount of blood drawn | 1 hour
  The total amount of blood drawn during the procedure
Number of attempts to place guidewire | 1 hour
  Number of attempts to place guidewire during the procedure
Arterial puncture rate | 1 hour
  The rate of arterial puncture during the procedure
Arterial puncture identification rate | 1 hour
  The rate of identification of arterial puncture
Success rate | 1 hour
  The rate for successful central venous catheterization within 3 attempts
Likert scale for satisfaction | 1 hour
  Likert scale for satisfaction of using either device for central venous catheterization and qualitative measurement for user experiences

CONTACTS AND LOCATIONS:
Overall Officials: Man-Ling Wang, MD, PhD, Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: The PI will review requests